CLINICAL TRIAL: NCT03100630
Title: An Open-label, Randomized, Parallel-group, Single Dose Study to Compare the Bioavailability of Subcutaneous Injections in the Arm, Thigh, and Abdomen and to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of RO7239361 in Healthy Participants
Brief Title: Compare Bioavailability of RO7239361 After Subcutaneous Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CN001-023; WP40225 (Other: Hoffman LaRoche Protocol ID)
Record Dates: First submitted 2017-03-29; First posted 2017-04-04 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A: RO7239361 (Active Comparator): RO7239361 subcutaneous injections on specified days; abdomen
  Interventions: Drug: RO7239361
- Treatment B: RO7239361 (Active Comparator): RO7239361 subcutaneous injections on specified days; arm
  Interventions: Drug: RO7239361
- Treatment C: RO7239361 (Active Comparator): RO7239361 subcutaneous injections on specified days; thigh
  Interventions: Drug: RO7239361

INTERVENTIONS:
Drug: RO7239361 — Specified dose on specified days

SUMMARY:
Randomized study in healthy men and women. Assess the similarity of RO7239361 when injected into the arm, thigh, or the stomach. Collect data on safety of RO7239361.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant as determined by no significant deviations in normal medical and surgical history and assessments
* Body Mass Index 18 kg/m2 to 32 kg/m2
* females must be of non-childbearing potential

Exclusion Criteria:

* tattoos or other skin findings on any of the potential injection sites
* history of chronic muscle pain within 30 days prior to study treatment
* prior history of IgG1 therapy

Other protocol defined inclusion and exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to 92 days
AUC from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to 92 days
AUC from time zero extrapolated to infinite time [AUC(INF)] | Up to 92 days

SECONDARY OUTCOMES:
Incidence of Adverse Events ( AEs) | Up to 92 days
Incidence of Serious Adverse Events (SAEs) | Up to 92 days
Change from baseline in electrocardiogram findings | Up to 92 days
Change from baseline in physical examination findings | Up to 92 days
Change from baseline in clinical laboratory test findings | Up to 92 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- WCCT Global, Inc., Cypress, California, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/